CLINICAL TRIAL: NCT07069452
Title: TARGET-ASPECT (Prognostic Value of Isolated and Combined Score Aspects in Acute Ischemic Stroke)
Brief Title: Prognostic Value of Isolated and Combined Score Aspects in Acute Ischemic Stroke
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0111_NEUROLOGIE
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Stroke, Ischemic; Thrombectomy; Thrombolytic Therapy; Brain Ischemia; Prognosis; Magnetic Resonance Imaging; Outcome Assessment (Health Care)
MeSH Terms: conditions — Ischemic Stroke; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study, called TARGET-ASPECT, looks at patients who had a type of stroke called acute ischemic stroke and were treated with clot-busting medicine and a procedure to remove the clot. Even with these treatments, about half of patients don't fully recover. The study aims to see if certain brain imaging scores, especially when combined, can better predict how well patients will recover 90 days after their stroke and if their blood vessels reopen successfully. The study will include 152 patients and last about 9 months. The goal is to find easy and reliable tools that doctors can use to make better treatment decisions.

ELIGIBILITY:
Inclusion Criteria :

* Patients aged 18 years or older
* Confirmed acute ischemic stroke on imaging
* Treated with both thrombolysis and thrombectomy
* Clinical follow-up data available at 90 days (mRS score)

Exclusion Criteria :

* Primary hemorrhagic stroke
* Early death or loss to follow-up without evaluation
* Poor-quality imaging that cannot be analyzed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 and over) who have experienced an acute ischemic stroke confirmed by imaging. These patients have undergone combined treatment with thrombolysis (clot-busting medication) and thrombectomy (mechanical clot removal). They are selected from a single medical center where detailed clinical and imaging follow-up data, including functional outcomes at 90 days, are available. Participants must have adequate-quality imaging and not have experienced early death or loss to follow-up before evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Favorable functional outcome defined as a mRS score of 0 to 2 at 90 days | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Gonesse, Gonesse, France